CLINICAL TRIAL: NCT04358393
Title: A Phase Ib/II Study of APG-115 Alone or in Combination With Azacitidine in Patients With Relapse/Refractory AML, CMML or MDS
Brief Title: A Study of APG-115 Alone or Combined With Azacitidine in Patients With AML, CMML, or MDS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APG115AU101
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: AML; Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; CMML; Myelodysplastic Syndromes; High-risk Myelodysplastic Syndrome; MDS
Keywords: TP53
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APG-115 monotherapy (Experimental): Monotherapy given in part 1
  Interventions: Drug: APG-115
- APG-115 + 5-azacitidine combination (Experimental): Combination therapy given in part 2
  Interventions: Drug: APG-115; Drug: 5-azacitidine

INTERVENTIONS:
Drug: APG-115 — APG-115 given once daily on day 1-5 of every 28 day cycle
Drug: 5-azacitidine — 5-AZA is given at 75 mg/m˄2/d subcutaneously daily on Day 1-7 every 28 days
  Other Names: Vidaza; Azadine
  Arms: APG-115 + 5-azacitidine combination

SUMMARY:
This is a two Part study in patients with relapsed/refractory acute myeloid leukemia (AML), chronic myelomonocytic leukemia (CMML), or high risk myelodysplastic syndrome (MDS) that will initially evaluate the safety and tolerability of APG-115 as a single agent in Part 1, followed by a combination of APG-115 + 5-azacitidine (5-AZA) in Part 2.

DETAILED DESCRIPTION:
Part 1: Dose escalation of APG-115 will use standard 3+3 design. APG-115 is administered orally once daily (QD) on Day 1-5 every 28-day cycle. The starting target dose is 100 mg (dose level; DL1) and will be increased in subsequent cohorts to 150 mg (DL2), 200 mg (DL3), and 250 mg (DL4), accordingly.

Part 2: Dose escalation of APG-115 in combination with 5-AZA will use standard 3+3 design. 5-AZA is administered at 75 mg/m˄2/d subcutaneously daily on Day 1-7 every 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of histologically confirmed relapsed or refractory AML, CMML, or high-risk MDS (overall revised international prognostic scoring system (IPSS-R) score > 3, including intermediate, high, or very high risk) by World Health Organization (WHO) classification for which no available standard therapies are indicated or anticipated to result in a durable response.
2. Adequate organ function as defined below:

   1. Liver function (total bilirubin < or = 1.5 x upper limit of normal (ULN), aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) <3 x ULN
   2. Kidney function (defined as a calculated creatinine clearance ≥ 60 mL/min; determined via urine collection for 24-hour creatinine clearance or by the Cockcroft Gault formula)
   3. Known cardiac ejection fraction of > or = 45% within the past 3 months
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
4. A negative serum pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
5. Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or legally authorized representative is required prior to their enrollment on the protocol.
6. Subject must have a projected life expectancy of at least 12 weeks.
7. Subject has a white blood cell count < 25 × 10˄9/L. Note: Hydroxyurea is permitted to meet this criteria.

Exclusion:

1. Pregnant women are excluded.
2. Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Have had leukemia therapy for 14 days prior to starting investigational drug. However, patients with rapidly proliferative disease may receive hydroxyurea as needed until 24 hours prior to starting therapy on this protocol and during the first cycle of study.
4. Have acute promyelocytic leukemia.
5. Active infection requiring systemic antibiotic/antifungal medication, known clinically active hepatitis B or C, or HIV infection.
6. Have received allogeneic hematopoietic stem cell transplant (HSCT) within 12 months prior to the first dose, or who have active/ongoing graft-versus host disease (GVHD), or require continued treatment with systemic immunosuppressive agents (calcineurin inhibitors within 4 weeks prior to the first dose), or received autologous hematopoietic stem cell transplantation within 6 months prior to the first dose.
7. Documented hypersensitivity to any of the components of the therapy program
8. Active, uncontrolled central nervous system (CNS) leukemia will not be eligible.
9. Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use at least 1 form of barrier birth control (such as condom) prior to study entry and for the duration of study participation.
10. Any prior systemic MDM2-p53 inhibitor treatment
11. Any other condition or circumstance that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.
12. History of other malignancies within 2 years prior to study entry, with the exception of:

    1. Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast
    2. Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin
    3. Previous malignancy confined and surgically resected (or treated with other modalities) with curative intention: requires discussion with sponsor
13. Failure to have recovered (Grade > 1) from prior treatment (including chemotherapy, targeted therapy, immunotherapy, experimental agents, radiation, or surgery)
14. Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block type II, 3rd degree block, or corrected QT interval (QTc) ≥470 msec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 28 days
  Part I is to assess the safety and tolerability of APG-115 by assessing the dose-limiting toxicity (DLT) of APG-115. End points include: Incidence of DLTs during the first 3 weeks of treatment of each dose cohort; Severity and frequency of any adverse event(s) (AE) and serious adverse event(s) (SAE) based on NCI CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Ascentage Pharma Group Inc.
Locations (8):
- United States (8):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Duke University, Durham, North Carolina
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - MD Anderson, Houston, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No